CLINICAL TRIAL: NCT05903989
Title: A Secondary Database Study Using COPD Cohort Study in Japan to Investigate Health Status of COPD Patients With Different Inhaler Treatment
Brief Title: Real-World Treatment Patterns and Patient Reported Outcome in COPD (REMIND)
Acronym: REMIND
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00080
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- LAMA
- LAMA plus LABA
- ICS plus LABA

SUMMARY:
This retrospective observational study aims to report distribution of the proportion of symptomatic Chronic obstructive pulmonary disease (COPD) patients classified by the COPD Assessment Test (CAT) managed with single or dual inhaler treatment using the data at cohort entry in the COPD cohort study, and treatment change and longitudinal CAT score by each inhaler treatment will also be evaluated using the data during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients taken with any of following inhaler treatments; LAMA, LAMA+LABA(both single and dual inhaler) or ICS+LABA(both single and dual inhaler) at cohort entry

Exclusion Criteria:

* Patients enrolled at the sites participated in the COPD cohort study where not agreed on secondary use of data for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out of 708 COPD patients registered in the COPD cohort study conducted in Japan, total of 448 patients received the following inhaler treatment at cohort entry will be included in this study; LAMA, LAMA+LABA or ICS+LABA .
  The patients not treated with the above-listed inhalers or with no COPD treatment at cohort entry will not be included for this study.
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with CAT (≥10, <10) at registration in each inhaler treatment group (Long acting muscarinic antagonist(LAMA), LAMA+Long acting β2 agonist(LABA) or Inhaled corticosteroid(ICS) +LABA) | At registration
  To describe the proportion of symptomatic(CAT ≥10) and non-symptomatic(CAT<10) COPD patients in each of 3 different inhaler treatment categories(LAMA, LAMA+LABA or ICS+LABA) at registration

SECONDARY OUTCOMES:
Proportion of patients with changes of inhaler treatment categories (step up or all other categories) during 1 year follow-up period by patients with CAT (≥10, <10) in each inhaler treatment group (LAMA, LAMA+LABA or ICS+LABA) at registration | 1 year follow-up
  To describe changes of inhaler treatment categories during the 1 year follow-up period in symptomatic/non-symptomatic COPD patients by 3 different inhaler treatment categories (LAMA, LAMA+LABA or ICS+LABA) at registration
Proportion of patients with all patterns of inhaler treatment category changes during 1 year follow-up period by patients with CAT (≥10, <10) in each inhaler treatment group (LAMA, LAMA+LABA or ICS+LABA) at registration | 1 year follow-up
  To describe changes of inhaler treatment categories during the 1 year follow-up period in symptomatic/non-symptomatic COPD patients by 3 different inhaler treatment categories (LAMA, LAMA+LABA or ICS+LABA) at registration
Proportion of patients with CAT (≥10, <10) after 1 year follow-up by patients with CAT (≥10, <10) in each inhaler treatment group (LAMA, LAMA+LABA or ICS+LABA) at registration | 1 year follow-up
  To describe the COPD symptom status assessed with CAT after 1 year follow-up period in symptomatic(CAT ≥10)/non-symptomatic(CAT<10) COPD patients by 3 different inhaler treatment categories (LAMA, LAMA+LABA or ICS+LABA) at registration
Mean change in the CAT scores between at registration and 1 year follow-up in each inhaler treatment group (LAMA, LAMA+LABA or ICS+LABA) at registration | 1 year follow-up
  To describe the change of COPD symptom status assessed with CAT during 1 year follow-up period by 3 different inhaler treatment categories (LAMA, LAMA+LABA or ICS+LABA) at registration

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Gon Y, Sorimachi R, Yoshida Y, Tamai Y, Takashima I, Arita Y, Sugiura H. Real-World Treatment Patterns and Patient-Reported Outcomes in Chronic Obstructive Pulmonary Disease in Japan: The REMIND Study. Adv Ther. 2024 Sep;41(9):3585-3597. doi: 10.1007/s12325-024-02927-5. Epub 2024 Jul 24. PMID 39046695
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00080&attachmentIdentifier=8f2c07c7-58d9-4a0c-8cdd-df719af59982&fileName=REMIND_Study_report_synopsis_v1.0.pdf&versionIdentifier=